CLINICAL TRIAL: NCT01164748
Title: Lymphatic Mapping After Previous Breast Surgery
Acronym: LABS
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Other Study IDs: NL22080.060.08
Record Dates: First submitted 2010-07-16; First posted 2010-07-19 (Estimated); Last update posted 2010-07-19 (Estimated); Status verified 2010-07

CONDITIONS: Breast Cancer; Sentinel Node
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Sentinel Node Biopsy: All women who has Sentinel Node Biopsy as their primary treatment of the axilla
  Interventions: Radiation: Lymphoscintigraphy
- Axillary Lymph Node Dissection: All women who had Axillary Lymph Node Dissection as primary axillary treatment
  Interventions: Radiation: Lymphoscintigraphy

INTERVENTIONS:
Radiation: Lymphoscintigraphy — in all women a lymphoscintigraphy was done to investigate drainage patterns of a previous operated breast and axilla
  Other Names: 99mTc-colloidal-albumin

SUMMARY:
Rationale: Like in primary breast cancer, prognosis in recurrent breast cancer is correlated with regional lymph node status. Therefore, axillary staging may be warranted in patients with recurrent disease and intact axillary nodes, although this has not been described in guidelines yet. The lymphatic drainage pathways in the breast and/or axilla could have been changed due to prior surgery and/or radiotherapy. These aberrant drainage pathways could be detected with lymphatic mapping and sentinel node biopsy (SNB), leading to a more accurate staging.

Objective: To assess the technical feasibility of lymphoscintigraphy after prior breast surgery. A second goal is to investigate whether or not previous breast surgery (with or without radiotherapy) significantly changes the lymphatic drainage pathways of the breast.

ELIGIBILITY:
Inclusion Criteria:

* treatment with BCT with SNB and/or ALND for primary breast cancer
* previous primary breast cancer located in the upper-outer quadrant of one breast
* Primary breast cancer treatment at least 3 years before the analysis, with or without adjuvant chemo- or hormonal therapy.

Exclusion Criteria:

* breast surgery for other reasons than breast cancer
* recurrent breast cancer
* former allergic reaction to 99mTc-colloidal albumin.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: We included patients that received BCT with SNB and/or ALND for primary breast cancer located in the upper-outer quadrant of one breast at least 3 years before this analysis. Patients were excluded if they had breast surgery for other reasons than breast cancer, had recurrent breast cancer or had a former allergic reaction to 99mTc-colloidal-albumin.
  44 patients were included and were divided into two groups according to previous surgical treatment of the axilla, being the sentinel node biopsy group and the Axillary Lymph Node Dissection group
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina Hospital, Eindhoven, Netherlands